CLINICAL TRIAL: NCT05979259
Title: Efficacy of a Digital School-Based Nutrition Education Intervention to Improve Children's Healthy Eating Knowledge, Attitudes and Behaviours
Brief Title: Examining the Impact of a Mobile Nutrition Education App for Child Nutrition Education in Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ontario Institute of Technology (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, JoAnne Arcand, Associate Professor, University of Ontario Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17109
Record Dates: First submitted 2023-07-13; First posted 2023-08-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Nutrition, Healthy
Keywords: Diet, Healthy; Digital Technology; Gamification; Health Education; School Health Services; Food Literacy
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Foodbot Factory) Group (Experimental)
  Interventions: Other: Serious game nutrition education intervention
- Control Group (Active Comparator)
  Interventions: Other: Conventional nutrition education intervention

INTERVENTIONS:
Other: Serious game nutrition education intervention — Classrooms will receive nutrition education lessons for 35-40 minutes for 5 consecutive days. As part of each lesson, students will play the "Foodbot Factory" nutrition education serious game for 10-15 minutes. The Foodbot Factory serious game and lessons are based on Ontario curriculum requirements and aligned Canada's Food Guide.
  Arms: Experimental (Foodbot Factory) Group
Other: Conventional nutrition education intervention — Classrooms will receive nutrition education lessons for 35-40 minutes for 5 consecutive days. As part of each lesson, students will use conventional learning activities, such as worksheets, sourced from an online teaching resource repository. The lessons are based on Ontario curriculum requirements and aligned Canada's Food Guide.
  Arms: Control Group

SUMMARY:
This trial will test the hypothesis that a digital curriculum-based nutrition education intervention using the Foodbot Factory serious game (i.e., a game designed for learning) leads to greater student engagement and learning about nutrition, compared to conventional nutrition education (e.g., worksheets), among students in Grades 4 and 5 in Ontario, Canada. This hypothesis is based on existing research suggesting that digital serious games, when well-integrated into the classroom setting, promote greater student engagement, learning and knowledge retention.

DETAILED DESCRIPTION:
This two-arm parallel cluster randomized controlled efficacy trial will determine if a digital curriculum-based nutrition education intervention (intervention group) leads to greater increases in overall nutrition knowledge compared to conventional nutrition education (control group) in Grade 4 and 4/5 classrooms after 1 week, and that it facilitates greater retention at 4 weeks and 3 months following the intervention period. Secondary outcomes include sub-scores of nutrition knowledge (i.e., knowledge of specific food groupings), nutrition attitudes, general child nutrition behaviours and dietary intakes. Due to the enhanced engagement serious games can provide, it is hypothesized that participants in the intervention group will show greater changes in and retention of their nutrition knowledge and nutrition behaviours. Thirty-two Grade 4 and 4/5 classrooms in Ontario, Canada will be randomized to the intervention or control group. Participants in both groups will receive nutrition education lessons for 35-40 minutes a day for five consecutive days. Participants in the intervention group will use the Foodbot Factory serious game while participants in the control group will use conventional learning materials (e.g., worksheets, teacher-led instruction). Both interventions will have these learning materials integrated into standardized nutrition education lesson plans. Overall and sub-scores of nutrition knowledge, and nutrition attitudes will be assessed using the Nutrition Attitudes and Knowledge questionnaire. General child nutrition behaviours (e.g., frequency of eating meals outside the home) will be assessed using a modified version of the Family Nutrition and Physical Activity Screening Tool and dietary intake will be assessed using the Block Food Screener for Ages 2-17. At baseline, parents and classroom teachers will respectively complete demographic questionnaires to measure co-variates that may impact outcomes of interest (e.g., household food security, presence of school food programs).

ELIGIBILITY:
Inclusion Criteria:

* Grade 4 or 4/5 classroom
* Classroom is located in a participating school board in Ontario

Exclusion Criteria:

* Classroom has already covered the "Healthy Eating" component of the Ontario Physical Health Education curriculum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Overall nutrition knowledge | Measured at baseline and immediately post-intervention (Day 5).
  Change in knowledge of healthy food choices based on Canada's Food Guide from baseline to immediately post-intervention as assessed by the Nutrition Attitudes and Knowledge Questionnaire. The minimum score is 0 and the maximum score is 20 with higher scores indicating higher knowledge.
Overall nutrition knowledge | Measured at baseline and 4 weeks post-intervention.
  Change in knowledge of healthy food choices based on Canada's Food Guide from baseline to immediately post-intervention as assessed by the Nutrition Attitudes and Knowledge Questionnaire. The minimum score is 0 and the maximum score is 20 with higher scores indicating higher knowledge.
Overall nutrition knowledge | Measured at baseline and 3 months post-intervention.
  Change in knowledge of healthy food choices based on Canada's Food Guide from baseline to immediately post-intervention as assessed by the Nutrition Attitudes and Knowledge Questionnaire. The minimum score is 0 and the maximum score is 20 with higher scores indicating higher knowledge.

SECONDARY OUTCOMES:
Drinks knowledge | Measured at baseline and immediately post-intervention (Day 5).
  Change in knowledge of drink choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Drinks knowledge | Measured at baseline and 4 weeks post-intervention.
  Change in knowledge of drink choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Drinks knowledge | Measured at baseline and 3 months post-intervention.
  Change in knowledge of drink choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Whole grain foods knowledge | Measured at baseline and immediately post-intervention (Day 5).
  Change in knowledge of whole grain food choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Whole grain foods knowledge | Measured at baseline and 4 weeks post-intervention.
  Change in knowledge of whole grain food choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Whole grain foods knowledge | Measured at baseline and 3 months post-intervention.
  Change in knowledge of whole grain food choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Vegetables & fruit knowledge | Measured at baseline and immediately post-intervention (Day 5).
  Change in knowledge of vegetable & fruit choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Vegetables & fruit knowledge | Measured at baseline and 4 weeks post-intervention.
  Change in knowledge of vegetable & fruit choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Vegetables & fruit knowledge | Measured at baseline and 3 months post-intervention.
  Change in knowledge of vegetable & fruit choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The maximum score on the scale is 5 with higher scores indicating higher knowledge.
Protein foods knowledge | Measured at baseline and immediately post-intervention (Day 5).
  Change in knowledge of protein food choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Protein foods knowledge | Measured at baseline and 4 weeks post-intervention.
  Change in knowledge of protein choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Protein foods knowledge | Measured at baseline and 3 months post-intervention.
  Change in knowledge of protein food choices based on Canada's Food Guide and assessed by the Nutrition Knowledge and Attitudes Questionnaire. The minimum score is 0 and the maximum score is 5 with higher scores indicating higher knowledge.
Nutrition attitudes | Measured at baseline and immediately post-intervention (Day 5).
  Change in attitudes towards nutrition and healthy eating assessed by the Nutrition Attitudes and Knowledge Questionnaire. Minimum score is 4 and maximum score is 20 with higher scores indicating more positive attitudes towards nutrition and healthy eating.
Nutrition attitudes | Measured at baseline and 4 weeks post-intervention.
  Change in attitudes towards nutrition and healthy eating assessed by the Nutrition Attitudes and Knowledge Questionnaire. Minimum score is 4 and maximum score is 20 with higher scores indicating more positive attitudes towards nutrition and healthy eating.
Nutrition attitudes | Measured at baseline and 3 months post-intervention.
  Change in attitudes towards nutrition and healthy eating assessed by the Nutrition Attitudes and Knowledge Questionnaire. Minimum score is 4 and maximum score is 20 with higher scores indicating more positive attitudes towards nutrition and healthy eating.
Dietary intake | Measured at baseline and immediately post-intervention (Day 5).
  Change in usual intake of foods (e.g., fruit, vegetables, whole grains), reported as average number of daily servings, over the past week assessed by the Block Food Screener Kids.
Dietary intake | Measured at baseline and 4 weeks post-intervention.
  Change in usual intake of foods (e.g., fruit, vegetables, whole grains), reported as average number of daily servings, over the past week assessed by the Block Food Screener Kids.
Dietary intake | Measured at baseline and 3 months post-intervention.
  Change in usual intake of foods (e.g., fruit, vegetables, whole grains), reported as average number of daily servings, over the past week assessed by the Block Food Screener Kids.
General nutrition behaviours | Measured at baseline and immediately post-intervention (Day 5).
  Change in behaviours relevant to nutrition and eating (e.g., frequency of consuming breakfast and meals outside the home) assessed by a modified version of the Family Nutrition and Physical Activity Screening Tool. There are 10 questions evaluating how often the child engages in a nutrition behaviour, with responses ranging from Never/Almost Never (1) to Very Often/Always (4). Changes in each behaviour will be reported independently.
General nutrition behaviours | Measured at baseline and 4 weeks post-intervention.
  Change in behaviours relevant to nutrition and eating (e.g., frequency of consuming breakfast and meals outside the home) assessed by a modified version of the Family Nutrition and Physical Activity Screening Tool. There are 10 questions evaluating how often the child engages in a nutrition behaviour, with responses ranging from Never/Almost Never (1) to Very Often/Always (4). Changes in each behaviour will be reported independently.
General nutrition behaviours | Measured at baseline and 3 months post-intervention.
  Change in behaviours relevant to nutrition and eating (e.g., frequency of consuming breakfast and meals outside the home) assessed by a modified version of the Family Nutrition and Physical Activity Screening Tool. There are 10 questions evaluating how often the child engages in a nutrition behaviour, with responses ranging from Never/Almost Never (1) to Very Often/Always (4). Changes in each behaviour will be reported independently.
Intervention acceptability | Measured immediately post-intervention (Day 5).
  Acceptability of the nutrition education interventions assessed by a questionnaire based on the Theoretical Framework of Acceptability. There are 11 questions evaluating different dimensions of intervention acceptability, with responses ranging from 1, indicating strong disagreement, to 5, indicating strong agreement (response options are specific to each question). Responses to each question will be reported independently.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Arcand, PhD, RD, Principal Investigator — University of Ontario Institute of Technology
Locations (1):
- University of Ontario Institute of Technology, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The research team aims to publish the study findings in a peer-reviewed journal and at academic conferences. The investigators will make an anonymized copy of the data available in an online repository.
Supporting Information: Study Protocol, SAP
Time Frame: When the study is complete, determined by the date on which the findings are published, electronic files will be stored for 5 years per guidelines from the Canadian Institutes of Health Research. Data can be made available following study completion, up until its disposal.
Access Criteria: Data will be made available to researchers upon reasonable request.

REFERENCES:
- [Background] Brown JM, Savaglio R, Watson G, Kaplansky A, LeSage A, Hughes J, Kapralos B, Arcand J. Optimizing Child Nutrition Education With the Foodbot Factory Mobile Health App: Formative Evaluation and Analysis. JMIR Form Res. 2020 Apr 17;4(4):e15534. doi: 10.2196/15534. PMID 32301743
- [Background] Froome HM, Townson C, Rhodes S, Franco-Arellano B, LeSage A, Savaglio R, Brown JM, Hughes J, Kapralos B, Arcand J. The Effectiveness of the Foodbot Factory Mobile Serious Game on Increasing Nutrition Knowledge in Children. Nutrients. 2020 Nov 6;12(11):3413. doi: 10.3390/nu12113413. PMID 33172094
- [Background] Franco-Arellano B, Brown JM, Froome HM, LeSage A, Arcand J. Development and pilot testing of the Nutrition Attitudes and Knowledge Questionnaire to measure changes of child nutrition knowledge related to the Canada's Food Guide. Appl Physiol Nutr Metab. 2021 Dec;46(12):1495-1501. doi: 10.1139/apnm-2021-0170. Epub 2021 Jul 21. PMID 34289315
- [Derived] Brown JM, Tahir S, Franco-Arellano B, LeSage A, Hughes J, Kapralos B, Lou W, Vogel E, Farkouh M, Tugault-Lafleur C, Arcand J. Efficacy of the Foodbot Factory digital curriculum-based nutrition education intervention in improving children's nutrition knowledge, attitudes and behaviours in elementary school classrooms: protocol for a cluster randomised controlled trial. BMJ Open. 2025 Jan 28;15(1):e092426. doi: 10.1136/bmjopen-2024-092426. PMID 39880422